CLINICAL TRIAL: NCT07355946
Title: The Effect of Nurse-Led Coaching Program on Self-Care Agency and Quality of Life in Reconstructed Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Sevil Güler, Professor Doctor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-77082166-302.08.01-1195604
Record Dates: First submitted 2025-12-28; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breast Reconstruction
Keywords: nursing; coaching; quality of life; self-care agency; Breast Reconstruction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data obtained from the intervention and control groups were coded as group one and group two in the SPSS program. During the statistical analysis of the data in the study, the intervention and control group data were masked, and the statistical analyses were performed by a different expert to ensure the statistician's blindness. The statistician had no information about which group the patients belonged to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention)
- Intervention Group (Experimental): A total of 9 sessions of nurse-led coaching program are implemented for the intervention group over 12 weeks.
  Interventions: Behavioral: Nurse-led Coaching Program

INTERVENTIONS:
Behavioral: Nurse-led Coaching Program — This intervention is implemented to increase patients' quality of life and self-care agency.
  Arms: Intervention Group

SUMMARY:
The primary objective of this clinical study is to examine the effects of a nurse-led coaching program on self-care agency in breast cancer patients who have undergone reconstruction. The secondary objective is to determine the opinions of patients who participated in the nurse-led coaching program for breast reconstruction surgery. Primary questions the study aims to answer are:

1. Is there a difference in self-care agency between breast reconstruction patients who received a nurse-led coaching program and those who did not?

   The secondary objective of this clinical study is to examine the effects of a nurse-led coaching program on quality of life in breast cancer patients who have undergone reconstruction. The secondary questions the study aims to answer are:
2. Is there a difference in quality of life between breast reconstruction patients who received a nurse-led coaching program and those who did not?

The researchers will compare whether there are differences in self-care agency and quality of life between breast cancer patients who received a nurse-led coaching program (intervention group) and those who did not (control group).

Participants:

* Patients who meet the inclusion criteria will be informed of the study's purpose during their postoperative hospital stay, and their informed consent will be obtained. Patients who agree to participate will complete an Introductory Information Form, the Self-Care Agency Scale, and the EORTC QLQ-C30 and QLQ-BR-42 Quality of Life Scales.
* After completing the pre-test measurements, the researchers will randomly assign patients to either the control or intervention groups using a random number table.
* Patients in the intervention group will receive a routine debriefing on the day of discharge and a total of nine coaching sessions, scheduled weekly for the first 6 weeks and biweekly for the following 6 weeks. These sessions will be conducted via online meeting.
* Patients in the control group will receive a routine debriefing only on the day of discharge.
* Post-test measurements will be administered to both groups at 12 weeks post-operatively.

DETAILED DESCRIPTION:
MATERIALS AND METHODS

1. Research Method This study was planned as a randomized controlled experimental study to determine the effects of a nurse-led coaching program on self-care agency and quality of life in breast cancer patients undergoing reconstruction.
2. Location and Characteristics of the Study The study is being conducted in 2025 at the Gazi University Health Research and Application Center (GUSAUM) Plastic Reconstructive and Hand Surgery Clinic and the Ankara Etlik City Hospital Plastic Surgery Clinic at Türkiye. In these clinics, breast reconstruction surgeries are performed simultaneously with breast cancer surgery, and in the early and late postoperative periods. Patients are admitted to the clinic the day before or on the day of surgery and undergo general anesthesia. Postoperative hospital stays are 1-3 days for patients undergoing breast reconstruction using breast implants, 3-4 days for patients undergoing TRAM flap reconstruction, and approximately 7-15 days for patients undergoing DIEP flap reconstruction. Apart from routine perioperative procedures, no special procedures are performed for breast reconstruction surgery at the clinic.

   Patients return to the outpatient clinic for follow-up visits 1-2 weeks after discharge and at one month. At three months postoperatively, the non-reconstructed breast is evaluated for equality with the reconstructed breast, and decisions are made about additional interventions. For patients undergoing core tissue breast reconstruction, the nipple and areola are also reconstructed during this process.
3. Research Universe and Sample Selection The research universe consisted of patients who underwent breast reconstruction due to breast cancer at GUSAUM Plastic, Reconstructive, and Hand Surgery and Ankara Etlik City Hospital Plastic Surgery Clinic.

   Inclusion criteria for the study were:
   * Patients who had undergone breast reconstruction surgery due to breast cancer,
   * Patients aged 18 and over,
   * Patients who understood and spoke Turkish,
   * Patients who agreed to participate voluntarily,
   * Patients who were literate.

   Exclusion criteria included:
   * Patients with speech, hearing, or visual impairments,
   * Patients with a psychiatric diagnosis or ongoing treatment,
   * Patients with metastatic breast cancer,
   * Patients with a cancer diagnosis other than breast cancer.

   The study termination criteria were:
   * Patients who wished to withdraw from the study during the follow-up period,
   * Patients who had a new cancer history during the follow-up period,
   * Patients who could not be reached when contacted five times in a row during the same week during the follow-up period,
   * Patients who did not regularly participate in the nurse-led coaching program (failing to attend three consecutive sessions or at least five total sessions),
   * Patients who died during the follow-up period.Implementation

   As a result of the power analysis conducted with the GPower 3.1.9.7 program, to determine the difference in self-care agency measurements between the groups, a sample size of 7 people was determined in each group, for a total of 14 people, based on Type 1 error: 0.05, Type 2 error: 0.20, and Effect Size = 1.636. However, due to differences in the structure of the study and the relatively low sample size, it was not deemed appropriate to use it as a reference. Taking into account the effect size ranges suggested by the program for cases where no similar studies exist, a sample size of 26 people was determined in each group, for a total of 52 people, based on Type 1 error: 0.05, Type 2 error: 0.20, and Effect Size = 0.80, to determine the difference in self-care agency and quality of life measurements between the groups. Taking into account the situation calculated due to possible losses in the study, the sample size was increased by 15%, and it was planned to include 60 people, 30 in each group.
4. Randomization and Blinding Simple randomization was used in the study. A random number table was used to randomly assign patients to the intervention and control groups. Because the patients in the intervention group were included in the coaching program, blinding of the patients in the study was not possible. Because the nurse-led coaching program was implemented by the researcher, researcher blinding was not possible. During the statistical analysis of the data in the study, the experimental and control group data will be masked, and the statistical analyses will be performed by a different expert, ensuring statistician blinding.
5. Data Collection Tools Data were collected using the Introductory Information Form, the Self-Care Agency Scale, and the EORTC QLQ-C30 and QLQ-BR42 Quality of Life Scales.

   5.1. Introductory Information Form The Introductory Information Form was developed by the researcher based on literature. This form contains a total of 24 questions regarding the individuals' sociodemographic characteristics (age, gender, height, weight, body mass index, marital status, cohabitants, education level, employment status, economic status, family history of breast cancer) and health status.

   5.2. Self-Care Agency Scale The Self-Care Agency Scale is a five-point Likert-type scale developed after the concept of self-care was introduced. The scale was developed by Kearney and Fleischer in 1979, and the first version consisted of 43 items. The Turkish version, whose validity and reliability study was conducted by Nahcivan in 1993, was revised to 35 items. Each statement on the scale is scored 0, 1, 2, 3, and 4, respectively. "Describes me a lot" receives 4 points, "Describes me a lot" receives 3 points, "I have no idea" receives 2 points, "Does not describe me" receives 1 point, and "Does not describe me at all" receives 0 points. Eight of the statements (3, 6, 9, 13, 19, 22, 26, and 31) are evaluated negatively, and the scoring is reversed. The highest score that can be obtained from the scale is 140, which represents the highest degree of self-care agency. In the Nahcivan study, Cronbach's alpha value was determined as 0.89.

   5.3. EORTC QLQ-C30 and QLQ-BR-42 Quality of Life Scales Developed by the European Organization for Research and Treatment of Cancer, EORTC, the EORTC QLQ-C30 Version 3.0 quality of life scale is a frequently used scale for cancer patients worldwide. The scale consists of 30 questions and three sub-items: general well-being, functional domain (physical function, role function, emotional function, cognitive function, social function), and symptoms (fatigue, nausea and vomiting, pain, shortness of breath, insomnia, loss of appetite, diarrhea, constipation, financial difficulties). The lowest possible score is 0, while the highest is 100. Questions 1-28 are on a four-point Likert-type scale, and questions 29 and 30 are on a seven-point Likert-type scale. Low scores on general well-being and functional domains indicate a decreased quality of life, while high scores indicate a higher quality of life. In the symptoms section, low scores indicate high quality of life, while high scores indicate low quality of life. The Turkish validity and reliability study of the scale was conducted by Beşer and Öz in 2003, and the Cronbach's alpha coefficient was found to be 0.82. The QLQ-BR42 is a continuation of the scale and consists of 42 questions investigating the side effects of breast cancer treatments, body image, sexuality, and future expectations. The scale's scoring is similar to the EORTC QLQ-C30 Version 3.0. Questions related to sexuality are reverse-scored. A high score on the functional domain and a low score on the symptoms section indicate a high quality of life. The validity and reliability study of the scale was conducted by Demirci and colleagues in 2011.
6. Application of the Research 6.1. Researcher Preparation To learn the art and competencies specific to the coaching profession, the researcher received two modules of training: 64 hours of theory and 16 hours of practical training from Anka Coaching, an institution accredited by the International Coach Federation (ICF) and the Association for Coaching (AC). As a result of these trainings, the researcher received the Art and Competencies of Coaching Certificate and the Holistic Life Coaching Certificate. At the end of the training, the researcher recorded one of her coaching sessions, which were listened to and evaluated by ICF mentors and deemed appropriate. As a result of this evaluation, the researcher was awarded the Holistic Coaching Certificate. The researcher developed her coaching skills by conducting voluntary coaching sessions. During the pre-implementation phase, the researcher conducted a total of six coaching sessions with two patients to gain experience in conducting coaching sessions with patients undergoing breast reconstruction surgery and to evaluate the effectiveness of the coaching program.

   6.2 Nurse-Led Coaching Program for Breast Reconstruction Patients The Nurse-Led Coaching Program for Breast Reconstruction Patients was developed by a researcher. The program includes literature review, the program's purpose, objectives, target audience, program flow, forms to be used in all coaching sessions, and coaching tools to be used when needed. Expert opinions were obtained from a total of nine experts regarding the Nurse-Led Coaching Program for Breast Reconstruction Patients. Three of the experts are MCC (Master Certified Coach - the highest-level title awarded to coaches) and are qualified in the field of coaching. The other experts are nursing academics who have also received coaching training and certification. A form was sent to the experts to provide their recommendations for all steps. The experts evaluated all sections of the program using a four-point Likert-type scale (1: not appropriate, 2: somewhat appropriate - major change needed, 3: appropriate - minor change needed, 4: very appropriate) and provided their recommendations on the prepared form. Based on expert opinions, the program's content validity ratio (CVR) was calculated using the Lawshe technique. The minimum value was determined as 0.75 based on the minimum values table for content validity ratios at a significance level of α=0.05 developed by Veneziano and Hooper. Analyses indicated that some sections of the program needed modifications. The coaching program was updated and revised based on feedback from the experts.

   The program's functionality was evaluated through a pre-implementation. As part of the Nurse-Led Coaching Program for Breast Reconstruction Patients, patients received coaching sessions for 12 weeks after discharge. There are differing opinions in the literature regarding the frequency and duration of coaching sessions. However, professional coaches trained by the International Coach Federation (ICF) and Association for Coaching (AC) recommend the frequency and duration of coaching sessions for each designated topic, three or four times a month, lasting approximately 35 minutes. Accordingly, a total of nine coaching sessions were conducted with the patients in the intervention group: weekly for the first 6 weeks after discharge and biweekly for the following 6 weeks. Each coaching session lasted an average of 30-40 minutes. Coaching sessions were conducted via online video calls using applications such as Zoom, WhatsApp, Skype, and Google Meets, as appropriate for the patient. In the first week, the nature of coaching was discussed with the patient, a coaching agreement was signed, and forms to assist with goal planning and agenda setting were introduced. In the second week, a Values Study for Breast Reconstruction Patients was conducted with the patient. In the third week, the Wheel of Life for Breast Reconstruction Patients was implemented, and in the fourth week, a SWOT Analysis for Breast Reconstruction Patients was conducted. In the following weeks, coaching sessions were conducted based on the agenda set by the patient. At the end of the coaching sessions, the patients were assessed for achievement of the goals they had set at the beginning of the session. A final counseling session was held 12 weeks after discharge, and the Wheel of Life was implemented again. The overall process and the effectiveness of the program were evaluated with the patient.
7. Data Evaluation The Statistical Package for Social Science (SPSS) 25.0 will be used for statistical analysis of the research data. Numbers, percentages, mean, and standard deviation values will be used to evaluate descriptive data. The Shapiro-Wilk test will assess compliance with a normal distribution. A t-test and a One-Way Analysis of Variance (ANOVA) for Repeated Measures will be used to compare the pretest and posttest mean scores of the intervention and control groups. A p value of <0.05 will be considered statistically significant. Intention-to-treat (ITT) analysis will be used for losses in the sample group during follow-up.
8. Ethical Aspects of the Research Permission for the study was obtained from the Gazi University Ethics Committee and the institutions where the study would be conducted. Written informed consent forms were signed by the patients participating in the study. Furthermore, the necessary permissions for the use of the data collection forms were obtained. After the study is concluded, patients in the control group will be contacted and voluntary coaching sessions (minimum 4 sessions) will be held for those who request it.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone breast reconstruction surgery due to breast cancer,
* Being 18 years of age or older,
* Being able to understand and speak Turkish,
* Voluntarily agreeing to participate in the study,
* Being able to read and write.

Exclusion Criteria:

* Having a speech, hearing, or vision impairment,
* Having a psychiatric diagnosis or ongoing treatment,
* Having metastatic breast cancer,
* Having a cancer diagnosis other than breast cancer.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 58 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Self-care Agency Scale | From enrollment to the end of coaching program at 12 weeks
  The Self-Care Agency Scale is a five-point Likert-type scale developed after the concept of self-care was introduced. The scale was developed by Kearney and Fleischer in 1979, and the first version consisted of 43 items (Kearney & Fleischer, 1979). The Turkish version, whose validity and reliability study was conducted by Nahcivan in 1993, was revised to 35 items. Each statement on the scale is scored 0, 1, 2, 3, and 4, respectively. "Describes me very much" receives 4 points, "Describes me very much" receives 3 points, "I have no idea" receives 2 points, "Does not describe me at all" receives 1 point, and "Does not describe me at all" receives 0 points. Eight of the statements (3, 6, 9, 13, 19, 22, 26, and 31) are evaluated negatively, and the scoring is reversed. The highest possible score on the scale is 140, representing the highest degree of self-care agency. In the Nahcivan study, Cronbach's alpha was determined to be 0.89.

SECONDARY OUTCOMES:
EORTC QLQ-C30 Quality of Life Scale | From enrollment to the end of coaching program at 12 weeks
  Developed by the European Organization for Research and Treatment of Cancer (EORTC) (2001), the EORTC QLQ-C30 Version 3.0 Quality of Life Scale is a frequently used measure for cancer patients worldwide. The scale consists of 30 questions and three sub-items: general well-being, functional domain and symptoms.

OTHER OUTCOMES:
EORTC QLQ-BR-42 Quality of Life Scale | From enrollment to the end of coaching program at 12 weeks
  Developed by the European Organization for Research and Treatment of Cancer (EORTC) (2001), the QLQ-BR42 is a continuation of the scale and consists of 42 questions investigating the side effects of breast cancer treatments, body image, sexuality, and future expectations. The scale's scoring is similar to the EORTC QLQ-C30 Version 3.0. Questions related to sexuality are reverse-scored. A high score on the functional domain and a low score on the symptoms section indicate a high quality of life.
Program Effectiveness Evaluation Form | At the end of the 12-week coaching program
  This form was created to evaluate the effectiveness of the program for participating patients. The form included three statements. Participants were asked to rate each statement on a scale of 1-10, from 1-Never to 10-Very. The first statement was: 'The coaching program increased my self-care ability.' The second statement was: 'The coaching program improved my quality of life.' The third statement was: 'I was satisfied with the coaching program.' The effectiveness of the program was evaluated by calculating the average and standard deviation of the scores given by the participants to these three statements.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Health, Research and Application Center, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data supporting this study are not publicly available due to ethical reasons but the datasets used and/or analyzed during the current study are available by emailing sevil.guler@gazi.edu.tr and nihalyildizemre@kku.edu.tr upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 2 years after the publication of results
Access Criteria: They will be able to access via e-mail to sevil.guler@gazi.edu.tr and nihalyildizemre@kku.edu.tr.